CLINICAL TRIAL: NCT01219491
Title: Do Egg Donor Recipient Characteristics Change Over Time?
Brief Title: Egg Donor Recipient Characteristics Preferences
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-00-16
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Egg Donor Recipient Characteristics
Keywords: egg donor; recipients; donor characteristics

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Egg donor recipients

SUMMARY:
To identify the characteristics in an egg donor that are important to a recipient and to see if those characteristics change over time.

DETAILED DESCRIPTION:
No study has explored how recipients' attitudes and reactions change over time regarding the selection criteria for their donors. Consequently, programs have no guidance in how to counsel prospective recipients as to whether their donor preferences will change over time. Participants will complete a survey at 4 points in time as they go through the process of selecting an egg donor and pursuing a pregnancy using that egg donor.

ELIGIBILITY:
All patients planning to undergo an egg donor cycle are eligible- there are no specific inclusion or exclusion criteria beyond that.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who are planning to undergo an egg donor cycle are eligible
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2007-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Characteristics of Donors | duration of study
  To identify the characteristics of donors which are important to recipients and whether their importance changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Braverman, PhD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (3):
- United States (3):
  - Reproductive Medicine Associates of Connecticut, Norwalk, Connecticut
  - Reproductive Medicine Assoicates of New Jersey, Morristown, New Jersey
  - Reproductive Medicine Associates of New York, New York, New York